CLINICAL TRIAL: NCT03895151
Title: Association Between Intakes of Protein, Calcium, and Milk With Gene Expression and Linear Growth of School Aged Children in Malang
Brief Title: Association Between Intakes of Protein, Calcium and Milk With Gene Expression and Linear Growth of School Aged Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SEAMEO Regional Centre for Food and Nutrition (Other)
Collaborators: Direktorat Riset dan Pengabdian Masyarakat Universitas Indonesia (Unknown); University of Brawijaya (Other)
Responsible Party: Principal Investigator, Dr.Umi Fahmida, Dr. Umi Fahmida, SEAMEO Regional Centre for Food and Nutrition
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NGMilkMalang
Record Dates: First submitted 2019-01-20; First posted 2019-03-29 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Nutritional Stunting; Nutritional Anemia; Nutritional Deficiency; Nutrigenetic; Nutrigenomic; Linear Programming; Food Based Recommendation
MeSH Terms: conditions — Malnutrition | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Milk supplementation (Experimental): Children will receive 130 ml fresh milk, 6 days/week for 20 weeks (January-June 2019).
  Milk will be provided and delivered by appointed supplier directly to school. Milk will be distributed with name of the student on the bottle - during break time.
  Subjects must be consumed with supervision of the teacher at school during the break.
  If they can not finish the milk at once, they can store it in the provided cool box. Student then can consume it again before they go home. Teacher have to record the remaining milk in each bottle that corresponds to every child name and record it in the provided form.
  Prior to holiday, student will be given the milk according to school leave days.
  Enumerators should collect the form every 3 days and make a recap in the provided form.
  Interventions: Dietary Supplement: Milk supplementation
- Food Based Recommendation (FBR) nutrition education (Experimental): FBR group will received nutrition education delivered by trained teacher under the supervision of researcher/research assistant once a week. Those who received nutrition education is not only the recruited subjects but also includes their classmates.
  Interventions: Other: Food Based Recommendation (FBR) nutrition education
- Control (No Intervention): Control group will receive standard nutrition education

INTERVENTIONS:
Dietary Supplement: Milk supplementation — Fresh milk from local farmer. No artificial sweetener and preservatives. Brandless.
  Arms: Milk supplementation
Other: Food Based Recommendation (FBR) nutrition education — Food Based Recommendation is result of OPTIFOOD WHO that analysed local food to optimize nutritional status according to problem nutrient.
  Arms: Food Based Recommendation (FBR) nutrition education

SUMMARY:
Protein is one type of nutrients known as the cause of stunting in developing countries since the mid-1970s (1) but then less attention on protein intake with the assumption that protein intake is sufficient. Compilation of published and non-published dietary intake research among Indonesian children aged 3-12 years (2), 0-18 years old (3) and 1-3 years old (3) found that protein intake among Indonesian children was sufficient (4). This finding is also confirmed by some other studies in 6 low-income countries and lead to the conclusion that growth restriction is not due to protein deficiency (5). Since then, micronutrient received main attention for the past 4 decades (1) to improve the health and survival of young children in developing countries. Issues on the need to re-examined protein recently emerge after the paper of Semba (1,6) regarding the low circulating amino acid among stunted children. It was hypothesized that the correlation between the low level of circulating amino acid with linear growth was through the mechanism of rapamycin complex C1 (mTORC1) and general control nonderepressible 2 (GCN2) pathway that contributes in the synthesis of sphingolipids and glycerophospholipids (6). However, the mechanism on how amino acid link to linear growth remains unclear.

Fortification among Asian children revealed that only milk as food vehicles reported a significant effect on linear growth (2). It is likely that the effect on linear growth is influenced not only on micronutrient content of the fortified foods but also on protein and amino acid profiles of milk as the food vehicle.

DETAILED DESCRIPTION:
Background:

The understanding of stunting has shifted from attention to protein and micronutrients in 60-80s to amino acids and calcium in the past two decades. Amino acids are suspected to be nutrients that determine to stunting because recent studies have shown that growth can be carried out by the information pathway through the mTOR pathway (the mechanistic target of rapamycin). mTOR is a serine/threonine protein kinase from the PI3K family related kinases which are the main subunits of 2 complex proteins, namely mTORC1 and mTORC2. The mTORC1 protein includes 5 main parts for cell growth, nutrition, growth factors, oxygen, energy, and stress. The mTORC2 protein is used in the cytoskeletal organization and cell survival. The activated mTORC1 protein initiates anabolic processes such as synthetic proteins, lipids, and nucleotides and inhibits catabolic processes such as autophagy. mTORC1 consists of three core proteins: mTOR, Raptor (regulatory protein associated with mTOR) and mLST8 (deadly mammals with Sec13 protein 8).

Activation of the mTORC1 pathway as a controller of growth and metabolism is in accordance with the adequacy of intracellular essential amino acids. Deficiency of leucine, isoleucine, and valine determines mTOR downregulation. Inadequate intake of essential amino acids will repress protein and lipid synthesis as well as cell growth that will affect bone and chondral palate growth, skeletal muscle growth, nervous system myelinization, immune function and the size of the organ formed (Saxton & Sabatini, 2017). Research by Semba, et.al (2016) shows that in stunting children's serum, the levels of the nine essential amino acids are very low. Given that the body does not form essential amino acids directly, the intake of amino acids from food becomes very important (Nuss & Tanumihardjo, 2011). Essential amino acids are mostly contained in animal protein, but consumption in developing countries is still limited. Consumption of animal food sources is associated with a lower risk of stunting.

Study of the mTORC1 pathway that has been done in vitro studies and experimental animals. In humans, the evidence of amino acid signaling through the mTORC1 pathway by using metabolomic aspects and proteomic and transcriptomic characteristics is still unknown. Analysis of genes related to MTORC1 pathway may answer this question

The scope of services:

1. To assess intakes of energy, macronutrients (protein, fat, carbohydrate), calcium and other micronutrients related to growth (zinc, iron, magnesium)
2. To assess linear growth
3. To assess gene expression of the mTORC1 pathway in school-age children in Malang, East Java.

The objective of research:

1. To assess energy and nutrient intake (especially for protein and calcium)
2. To assess the expression of mTOR gene
3. To assess the linear growth (height)
4. To assess the association between intake of protein, calcium, milk with gene expression of mTOR and linear growth of children who received food-based intervention with or without milk with comparable calcium and protein intakes

ELIGIBILITY:
Inclusion Criteria:

* Primary school children
* Willing to take part in the research and taken venous blood sampling as evidence by the signing of an informed consent from the parents
* Does not suffer from disability
* No complaint such as diarrhea, vomiting or nausea after drinking milk (based on the information of parents during screening)

Exclusion Criteria:

* The child not present when taking blood
* Having a history of bleeding such as hemophilia
* Children have plans to move schools within the next 6 months from the baseline data collection.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Increasing of children height who receive intervention from baseline | 3 days in end-line of study
  Height of the subject will be measured using Shorrboard. Height measurement will be taken twice, the difference between 1st and 2nd measurements should be not more than 0.7 cm. The data analyzed using WHO AnthroPlus to obtain height for age z-score (HAZ) of the subject.

SECONDARY OUTCOMES:
nutrient intakes | 3 days in baseline and end-line
  Dietary of energy intake, macronutrients, calcium and other micronutrients related to growth will be assessed using 24-hour recall with multiple-pass interviewing technique. The analysis will be performed using Nutrisurvey 2017 with Indonesian food composition table.
VDR Gene Polymorphism of SNP rs4516035 and rs11568820 | in middle of study (2 months after baseline)
  The SNP Genotyping assay analyzed using Real Time PCR and StepOne V2.3 Software. A total of 40 cycles will performed. The cycling steps of the analysis are Hold (95oC, 20s), Denaturation (95oC, 3s), Annealing Extension (60oC, 20s). The total running time was about one and a half hours for 40 cycles.
gene expression of mTORC1 pathway | 3 days in end-line of study
  The expression of 5' TOP genes as biomarker of downstream mTORC1 pathway will be analyzed using RT-qPCR and StepOne V2.3 Software. mRNA quantified by SYBR Green reaction. A total of 40 cycles will performed. The cycling steps of the analysis are UDG activation (50oC, 2min), Dual-Lock DNA polymerase (95oC, 2min), Denaturation (95oC, 3s), Annealing Extension (60oC, 30s). The total running time was about half an hour for 40 cycles.

CONTACTS AND LOCATIONS:
Overall Officials: Umi Fahmida Fahmida, Dr, Principal Investigator — SEAMEO RECFON
Locations (1):
- Universitas Brawijaya, Malang, East Java, Indonesia